CLINICAL TRIAL: NCT00164905
Title: Role of Doppler Ultrasound in Severe Peptic Ulcer Hemorrhage: Can it Guide the Use of and Predict Failure of Endoscopic Treatment? A Prospective, Multicenter, Randomized, Controlled Study
Brief Title: Role of Doppler Ultrasound in Severe Peptic Ulcer Hemorrhage
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DOP-US study
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: Peptic ulcer hemorrhage; Doppler ultrasound
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doppler ultrasound (Active Comparator)
  Interventions: Device: Doppler ultrasound probe
- No Doppler ultrasound (No Intervention)

INTERVENTIONS:
Device: Doppler ultrasound probe — Applying to ulcer base to assess the blood flow underneath the ulcer
  Other Names: DOP_US
  Arms: Doppler ultrasound

SUMMARY:
The aim of study is to evaluate whether Doppler ultrasound can accurately identify patients who are at risk of recurrent bleeding, who will require endoscopic therapy, and who will fail endoscopic therapy.

DETAILED DESCRIPTION:
Bleeding peptic ulcer is a life-threatening emergency. Endoscopic therapy is a proven technique in the acute hemostasis of bleeding ulcers. Currently there is no objective assessment of adequacy of endoscopic therapy. Endoscopic Doppler ultrasound enables endoscopists in detecting blood flow in a vessel beneath an ulcer. A persistent signal after endoscopic therapy predicts recurrent bleeding. The current study proposes to compare assessment of ulcer base using either Doppler ultrasound or endoscopists' interpretation of ulcer floors. The trial design is one of a prospective randomized controlled cross-over study in which patients with severe upper gastrointestinal bleeding and documented peptic ulcers at endoscopy are enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Clean base ulcer with severe upper GIB (defined as melaena, hematochezia, hematemesis, and/or gross blood in NG lavage), and any one of the following:

  1. SBP ≤ 90mmHg; P of ≥110 bpm; or orthostatic changes with SBP drops 20mmHg or P increases 20 bpm; or,
  2. Transfusion of 2 or more units of packed red blood cells within 12 hrs of admission; or,
  3. A documented HCT drop of at lest 6% from baseline.
* Endoscopically confirmed bleeding from GU, DU, pyloric ulcer, or anastomotic ulcer
* Pt can either have primary or secondary acute UGI haemorrhage

Exclusion Criteria:

* Bleeding site from lesion other than GU, DU, pyloric or anastomotic ulcer
* there is more than one type of significant bleeding lesion
* Documented hx of cirrhosis / portal HT
* ESRF requiring any form of dialysis
* Expected or persistent (>24hrs) coagulopathy with INR> 1.5
* Platelet count is under 50000/mm3
* Aspirin User / Plavix [Clopidogrel] User
* If the ulcer is neoplastic
* Cannot obtained consent
* Age < 18 or is pregnant
* Severe comorbid of which life expectancy <30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2004-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Recurrent bleeding | Within 30 days

SECONDARY OUTCOMES:
Length of stay | Within 56 days
ICU utilization | Within 56 days
Blood Transfusion during hospital | Within 56 days
Need for urgent/emergent ulcer surgery for bleeding | Within 56 days
Need for angiographic treatment of bleeding | Within 56 days
Death | within 56 days

CONTACTS AND LOCATIONS:
Overall Officials: James Y Lau, MD, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong SAR, China